CLINICAL TRIAL: NCT00980967
Title: Predictive Factors for Chronic Rejection in Lung Transplant Recipients: COLT Study
Acronym: COLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: CHU de Nantes, CHU de Nantes
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BRD 09/1-F
Record Dates: First submitted 2009-09-11; First posted 2009-09-21 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Rejection; Lung Transplantation
Keywords: Lung transplantation; Chronic lung rejection; Obliterative bronchiolitis; Predictive factors
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Study of predictive factors — Identification of predictive factors for lung chronic rejection outcome in lung transplant recipients

SUMMARY:
Obliterative Bronchiolitis (OB) is the major cause of long-term lung allograft loss for patients with end stage pulmonary diseases like cystic fibrosis. Numerous cells and proteins are implicated in this process, which have never been studied prospectively in a multicentric longitudinal cohort. The aim of this study is to detect predictive risk factors of OB through a national multicentric cohort of 500 newly transplanted recipients (COLT). COLT will consist in a large database, associated with a recipient bio-collection, and specific projects using these resources. COLT will aggregate all the 11 French centres of pulmonary transplantation. Patient will be followed-up during 5 years. Blood samples will be obtained. Induced sputum, bronchoalveolar lavage fuid, exhaled breath condensate and trans bronchial biopsies will be also taken. T cells, known to be involved in chronic rejection will be studied, and genomic, microarray and proteomic approaches will be used to detect further predictive factors. A study on Circulating Endothelial Cells and Circulating Endothelial Progenitors is also realised from blood samples. COLT will prove molecular markers to be predictive of early OB, before the development of severe airway obstruction and will allow the identification of patients at high risk of OB. COLT will identify potential targets for future treatments of OB. This collaborative project makes research and clinical teams working together, and creates the conditions of a long term network, extendable to other laboratories with new projects and additional European transplant centres.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥ 18 years
* who have signed an Inform Consent Form
* double or heart-lung transplant recipients

Exclusion Criteria:

* Pregnant or nursing women
* Patients with concomitant chronic inflammatory disease, independently of acute or chronic rejection or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2009-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive factors for lung chronic rejection outcome in lung transplant recipients. This primary outcome will be evaluated at the end of the study. | 8 years

SECONDARY OUTCOMES:
Evaluate the pertinence of a monitoring of lung chronic rejection based on the predictive factors identified in the study, in order to prevent this rejection. The secondary outcome measure will be evaluated at the end of the study. | 8 years

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU de Bordeaux, Bordeaux
  - CHU de Grenoble, Grenoble
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - CHU de Lyon, Lyon
  - CHU de Marseille, Marseille
  - CHU Nantes, Nantes
  - HEGP, Paris
  - Hôpital Bichat, Paris
  - CHRU de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Reucherand B, Tissot A, Lacoste P, Roux A, Coiffard B, Demant X, Magnan A, Renaud-Picard B, Le Pavec J, Merveilleux C, Villeneuve T, Falque L, Salpin M, Carlier N, Knoop C, Reynaud-Gaubert M, Kessler R, Dauriat G, Lair D, Nieves A, Foucher Y, Roussel JC, Senage T; COLT Consortium. Effect of Donor Age on Survival in Lung Transplantation: A Multicentric Retrospective Study. Eur J Cardiothorac Surg. 2025 Dec 1;67(12):ezaf420. doi: 10.1093/ejcts/ezaf420. PMID 41432731
- [Derived] Brugiere O, Dreyfuss D, Guilet R, Rong S, Hirschi S, Renaud-Picard B, Reynaud-Gaubert M, Coiffard B, Bunel V, Messika J, Demant X, Le Pavec J, Dauriat G, Saint Raymond C, Falque L, Mornex JF, Tissot A, Lair D, Le Borgne Krams A, Bousseau V, Magnan A, Picard C, Roux A, Glorion M, Carmagnat M, Gazeau F, Aubertin K, Carosella E, Vallee A, Landais C, Rouas-Freiss N, LeMaoult J; the COLT Consortium. Circulating Vesicular-bound HLA-G as Noninvasive Predictive Biomarker of CLAD After Lung Transplantation. Transplantation. 2025 Apr 1;109(4):736-745. doi: 10.1097/TP.0000000000005175. Epub 2024 Sep 19. PMID 39294868
- [Derived] Durand M, Lacoste P, Danger R, Jacquemont L, Brosseau C, Durand E, Tilly G, Loy J, Foureau A, Royer PJ, Tissot A, Roux A, Reynaud-Gaubert M, Kessler R, Mussot S, Dromer C, Brugiere O, Mornex JF, Guillemain R, Claustre J, Degauque N, Magnan A, Brouard S; COLT and SysCLAD Consortia. High circulating CD4+CD25hiFOXP3+ T-cell sub-population early after lung transplantation is associated with development of bronchiolitis obliterans syndrome. J Heart Lung Transplant. 2018 Jun;37(6):770-781. doi: 10.1016/j.healun.2018.01.1306. Epub 2018 Mar 20. PMID 29571601
- [Derived] Benmerad M, Slama R, Botturi K, Claustre J, Roux A, Sage E, Reynaud-Gaubert M, Gomez C, Kessler R, Brugiere O, Mornex JF, Mussot S, Dahan M, Boussaud V, Danner-Boucher I, Dromer C, Knoop C, Auffray A, Lepeule J, Malherbe L, Meleux F, Nicod L, Magnan A, Pison C, Siroux V; SysCLAD consortium. Chronic effects of air pollution on lung function after lung transplantation in the Systems prediction of Chronic Lung Allograft Dysfunction (SysCLAD) study. Eur Respir J. 2017 Jan 18;49(1):1600206. doi: 10.1183/13993003.00206-2016. Print 2017 Jan. PMID 28100545
- [Derived] Pison C, Magnan A, Botturi K, Seve M, Brouard S, Marsland BJ, Ernst F, Paprotka T, Deplanche K, Fritz A, Siroux V, Boissel JP, Corris PA, Auffray C, Nicod LP; SysCLAD consortium. Prediction of chronic lung allograft dysfunction: a systems medicine challenge. Eur Respir J. 2014 Mar;43(3):689-93. doi: 10.1183/09031936.00161313. No abstract available. PMID 24585866